CLINICAL TRIAL: NCT00250198
Title: A Randomized, Double-blind, Pilot Study of the Oral IL-12/23 Inhibitor, STA-5326 Mesylate, to Investigate Peripheral Blood and Mucosal Mononuclear Cell Phenotype and Cytokine Responses in Patients With Crohn's Disease
Brief Title: The Immunological and Blood Effects of STA-5326 Mesylate on Patients With Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 060021; 06-I-0021
Record Dates: First submitted 2005-11-05; First posted 2005-11-07 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2006-09-05

CONDITIONS: Crohn's Disease
Keywords: T Cell; Lymphocyte; Lamina Propria; Colonoscopy; Placebo; Crohn's Disease; Crohns Disease
MeSH Terms: conditions — Crohn Disease | interventions — apilimod

INTERVENTIONS:
Drug: STA-5326

SUMMARY:
This study will test whether a new experimental drug called STA-5326 mesylate will decrease inflammatory chemicals called cytokines in patients with Crohn's disease. The drug has prevented gut inflammation in mice and rats and has improved symptoms in humans with active Crohn's disease.

Patients with Crohn's Disease between 18 and 75 years of age and who have active disease symptoms may be eligible for this study. Candidates are screened with a review of their medical records, a medical history and physical examination, electrocardiogram, blood and urine tests, chest x-ray and tuberculin skin test. They fill out diary cards for 7 days (measuring their symptoms on the Crohn's Disease Activity Index, or CDAI) and complete a 32-item Inflammatory Bowel Disease Questionnaire (IBDQ) that surveys how their disease affects their live and activities.

Participants have a colonoscopy (an examination of the colon using a lighted tube) before starting the study medication. Colon tissue samples are biopsied during the procedure. Following the colonoscopy, patients are randomly assigned to receive either STA-5326 mesylate or placebo (sugar or dummy pill). They take four tablets a day and are seen in the clinic once a week (days 1, 8, 15, 22 and 29) for the following tests and procedures:

* Physical examination - Days 1, 8, 15, 22, 29
* Blood tests - Days 1, 8, 15, 22, 29
* Pharmacodynamic study (blood collected before the first dose of medicine and again after 1, 2, 4, 6 and 8 hours to measure levels of the drug in the blood) - Day 1
* CDAI and IBDQ - Days 1, 15, 29
* Review of medications and symptoms - Days 1, 8, 15, 22, 29
* EKG - Days 8, 29
* Pregnancy test for women of child-bearing potential - Days 15, 29
* Urine test - Day 29

After patients complete the above treatment and tests, they undergo a second colonoscopy within 48 hours of their last dose of study medication and may be offered another 1-week supply of medication. Those for whom additional treatment is deemed potentially beneficial are offered another 4-week course of drug or placebo (continuing whichever they took the first 4 weeks). They come to the clinic for two visits 2 weeks apart (days 43 and 57) for a physical examination, blood tests, EKG, pregnancy test for women, CDAI, IBDQ and review of medications and symptoms. A urine sample is collected only on day 57. A third colonoscopy is done after all the tests are completed on day 57, within 48 hours after the last dose of study medication.

Patients return to the clinic about 1 week after their final dose of study medication (day 36 for patients who complete only 1 month of treatment and day 64 for those who complete a second month of treatment) for a limited physical examination, blood tests, pregnancy test for women, CDAI and IBDQ, and a review of their medications and symptoms.

DETAILED DESCRIPTION:
The purpose of this study is to measure the mucosal immunological effects and peripheral blood effects of the oral IL-12/23 inhibitor, STA-5326 mesylate, in subjects with active Crohn's disease (CD). Crohn's disease is a chronic, relapsing inflammatory condition of the small and large bowel associated with excessive Th1 cytokine production. Since IL-12 is a key cytokine driving the Th1 response, novel therapies targeting IL-12 have been successful in treating CD in animal models and in humans. Data from humans and from animal models further suggest that both IL-12 and IL-23 may have a role in this active gut inflammation. STA-5326 mesylate is an oral drug that suppresses IL-12p40 production (a subunit shared by IL-12 and IL-23) in vitro and has apparent safety and clinical activity in a recent open-label trial of treatment for CD.

This protocol will enroll and randomize 12 subjects with moderate to severe active CD (CD Activity Index [CDAI] 220 to 450, inclusive) for 4 weeks of daily study drug treatment (9 subjects will receive 100 mg STA-5326 mesylate and 3 will receive placebo). Subjects will be evaluated for safety that will include monitoring of adverse events and concomitant medications, clinical laboratory testing, electrocardiogram (ECG) tracings, and physical examinations including vital signs. Efficacy assessments will include the CDAI, the Simple Endoscopic Score for CD (SES-CD), results from the Inflammatory Bowel Disease Questionnaire (IBDQ), and changes from Baseline for plasma C reactive protein (CRP) (measured by high sensitivity assay). In addition, immunologic effects (lymphocyte phenotyping cytokine secretion from peripheral blood and lamina propria mononuclear cells [LPMCs]) will be assessed. Descriptive statistics (n, mean, median, standard deviation, minimum and maximum range) will be used to summarize data for each treatment group.

ELIGIBILITY:
* INCLUSION CRITERIA:

A subject is eligible for the study if all of the following criteria are met:

Has given written informed consent prior to Screening.

Is male or female aged 18 through 75 years.

Has CD diagnosed definitively prior to Screening (based upon clinical, endoscopic, radiologic imaging, or histological assessments).

Has a CDAI score of 220 to 450, inclusive.

If taking sulfasalazine or mesalamine, must have been using continuously for at least 2 months prior to randomization and at stable doses for at least 2 weeks prior to randomization.

If taking azathioprine, 6-mercaptopurine, or methotrexate, must have used continuously for at least 3 months prior to randomization and at stable doses for at least 1 month prior to randomization.

If taking oral antibiotics chronically, must have used continuously for at least 1 month prior to randomization and at stable doses for at least two weeks prior to randomization.

If taking corticosteroids, must be taking prednisone less than or equal to 20 mg daily (or equivalent), or budesonide less than or equal to 9 mg daily for at least 2 months prior to randomization and at stable doses for at least 2 weeks prior to randomization.

Not taking any potential CYP3A4 inhibitors/inducers (eg, macrolide antibiotics, HIV protease inhibitors, antifungals, grapefruit juice, St. John's Wort).

EXCLUSION CRITERIA:

A subject is excluded from the study if any of the following criteria are met:

General criteria:

Has any clinically significant disease (eg, renal, hepatic, neurological, cardiovascular, pulmonary, endocrinologic, psychiatric, hematologic, urologic, or other acute or chronic illness) that in the opinion of the investigator would make the subject an unsuitable candidate for this trial.

Is a woman who has a positive pregnancy test or who is breast-feeding

Is a woman of childbearing potential or a man who does not agree to use 2 forms of contraception during the course of the study and Follow-up period.

Has hypersensitivity to any of the components of STA 5326 mesylate drug product.

Has any of the following clinical chemistry values:

* AST greater than 2.0 x ULN.
* ALT greater than 2.0 x ULN.
* Serum bilirubin greater than 1.5 x ULN.
* Serum creatinine greater than 1.5 x ULN.
* Alkaline phosphatase greater than 2.5 x ULN.

Has a hemoglobin level less than 9 g/dL or hematocrit less than 30%.

Has a PT INR greater than 1.3 or PTT of 3 or more seconds longer than control values.

Has the following cell counts (cells/microliter):

* Platelets less than 100,000 or greater than 800,000.
* White blood count less than 3,500.
* Neutrophils less than 2000.

Has a history of any infection requiring intravenous antibiotics, a serious local infection (eg, cellulitis, abscess) or systemic infection (eg, pneumonia, septicemia) that occurred within 3 months of randomization.

Has a history of cancer within the past 5 years, with the exception of excised basal cell carcinoma, squamous cell carcinoma of the skin, or cervical carcinoma in situ.

Had a dependency for any illicit drug, chemical, or alcohol within the past 5 years.

Has a history of active tuberculosis, a positive PPD skin test, acute or chronic hepatitis B, hepatitis C, or human immunodeficiency virus (HIV).

Gastrointestinal criteria:

Has a current ileostomy or colostomy.

Has a proctocolectomy or total colectomy.

Has short bowel syndrome requiring enteral or parenteral nutrition supplementation or total parenteral nutrition.

Has a stool sample positive for gastrointestinal infection (eg, Clostridium difficile toxin, etc.) during Screening.

Has a history or diagnosis of ulcerative or indeterminate colitis.

Had bowel surgery in the previous 3 months.

Had severe intestinal tract stenosis or fixed strictures causing symptomatic obstruction within 6 months prior to randomization.

Prior medication criteria relative to randomization:

Received parenteral corticosteroids or corticotropin within 1 month prior to randomization.

Has had regular use of aspirin or other non-steroidal anti-inflammatory drugs within 2 weeks prior to randomization (other than use of chronic low dose aspirin [81 mg per day] for cardioprotective effects).

Received any investigational drug within 3 months prior to randomization.

Received cyclosporine, tacrolimus, sirolimus, or mycophenolate mofetil within 2 months prior to randomization.

Received any biological product (eg, infliximab, adalimumab, natalizumab, etc.) within 3 months prior to randomization.

Ever received treatment with STA-5326 mesylate, IL-12 antibodies, or other specific IL-12 inhibitors.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12
Dates: Start 2005-11-03; Study Completion 2006-09-05

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Allergy and Infectious Diseases (NIAID), Bethesda, Maryland, United States

REFERENCES:
- [Background] Larsson S, Linden M. Effects of a corticosteroid, budesonide, on production of bioactive IL-12 by human monocytes. Cytokine. 1998 Oct;10(10):786-9. doi: 10.1006/cyto.1998.0362. PMID 9811532